CLINICAL TRIAL: NCT04039945
Title: Fr1da Early Diagnosis and Care of Type 1 Diabetes
Acronym: Fr1da
Status: Recruiting | Type: Observational
Sponsor: Helmholtz Zentrum München (Industry)
Responsible Party: Principal Investigator, Anette-Gabriele Ziegler, Prof. Dr.med. Anette-G. Ziegler, Director, Institute of Diabetes Research, Helmholtz Zentrum München
Other Study IDs: 808040014
Record Dates: First submitted 2019-07-26; First posted 2019-07-31 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Fr1da; Fr1da-Plus; type 1 diabetes; islet autoantibodies
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Fr1da study: "Early diagnosis and care of type 1 diabetes" aims to carry out a comprehensive, population-based screening for the early diagnosis of type 1 diabetes as part of the U7 to U11 preventive medical check-up for children or between the ages of 2 and 10 years in Bavaria and to implement it in other federal states. Screening is recommended at two time points: 1st screening at the age of 3 years (U7a) and 2nd screening at the age of 7 years (U10). In addition, relatives of patients with type 1 diabetes between the ages of 1 and 21 can be screened repeatedly at intervals of 3 to 5 years for an early-stage of type 1 diabetes.

DETAILED DESCRIPTION:
With the Fr1da study, 100,000 children in the Free State of Bavaria were offered a one-off screening for the early diagnosis of type 1 diabetes from January 1, 2015 to 2019 as part of the U7 (21st month of life) to U9 (64th month of life) check-ups, or as part of any other visit at the paediatrician between the ages of 2 and 5. After 100,000 children had been screened in the Fr1da study, the screening was continued as part of Fr1da (formerly Fr1da-Plus). The screening was then extended to a second age group from 6 to 10 years (U10-U11). As relatives of people with type 1 diabetes have an up to 10-fold increased risk of developing type 1 diabetes themselves, the screening is also offered to these people between the age 1 to 21 years. The aim of the Fr1da study is 1) to prevent life-threatening ketoacidosis at clinical manifestation of type 1 diabetes, 2) to reduce anxiety, uncertainty and psychological stress through training and intensive support for those affected, 3) to test the feasibility of two-time nationwide screening and evaluate the benefits, 4) to determine the prevalence of early-stage type 1 diabetes in children in defined age groups and in first and second screening, 5) to identify geographical differences and associations with environmental factors in the development and progression of the disease and 6) to prevent disease progression by means of preventive therapies. From 2024, the screening will also be offered in other federal states outside of Bavaria.

ELIGIBILITY:
written informed consent by one custodial parent

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children between the ages of 2 and 10 years
Sampling Method: Non-Probability Sample
Enrollment: 285000 (Estimated)
Dates: Start 2015-02 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
presence of multiple islet autoantibodies | up to 3 years
  multiple islet autoantibodies (IAA, GADA, IA-2A and/or ZnT8A)

CONTACTS AND LOCATIONS:
Locations (1):
- Institut für Diabetesforschung, Helmholtz Zentrum München, Munich, Germany

REFERENCES:
- [Derived] Hippich M, Holthaus L, Assfalg R, Zapardiel-Gonzalo J, Kapfelsperger H, Heigermoser M, Haupt F, Ewald DA, Welzhofer TC, Marcus BA, Heck S, Koelln A, Stock J, Voss F, Secchi M, Piemonti L, de la Rosa K, Protzer U, Boehmer M, Achenbach P, Lampasona V, Bonifacio E, Ziegler AG. A Public Health Antibody Screening Indicates a 6-Fold Higher SARS-CoV-2 Exposure Rate than Reported Cases in Children. Med. 2021 Feb 12;2(2):149-163.e4. doi: 10.1016/j.medj.2020.10.003. Epub 2020 Oct 29. PMID 33163984